CLINICAL TRIAL: NCT01081808
Title: A Phase I Study of Anti-CD3 x Cetuximab-Armed Activated T Cells, Low Dose IL-2, and GM-CSF for EGFR-Positive, Advanced Solid Tumors
Brief Title: Laboratory-Treated Autologous Lymphocytes, Aldesleukin, and Sargramostim (GM-CSF) in Treating Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Roger Williams Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RWH 111-32
Record Dates: First submitted 2010-01-28; First posted 2010-03-05 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Neoplasms; Tumors; Solid Tumors; Metastatic Cancer
Keywords: PhaseI; Solid Tumor; biomarkers; T cell; Cetuximab; Epidermal Growth Factor Receptor; Aldesleukin; Lymphocytes; Autologous; Recurrent; Refractory; Metastatic; Immunotherapy; Antibodies; Neoplasms by Site; Anti-Retroviral Agents; Therapeutic Uses; Anti-Infective Agents; Neoplasms by Histologic Type; Antineoplastic Agents; Antiviral Agents; Pharmacologic Actions; Carcinoma; Neoplasms
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Recurrence; Neoplasms by Site; Neoplasms by Histologic Type; Carcinoma | interventions — Interleukin-2; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Armed Activated T Cells (Other): Activated T Cells (ATC) armed with the bispecific antibody OKT3 x Cetuximab (EGFRBi). ATC will be expanded for 14 days from a leukapheresis product, armed with EGFRBi, cryopreserved and infused in 8 divided doses. Patients will also receive low dose subcutaneous IL-2(3000,000 IU/m2/day) and GM-CSF (250ug/m2 twice per week)
  Interventions: Biological: EGFRBi-armed autologous activated T cells

INTERVENTIONS:
Biological: EGFRBi-armed autologous activated T cells — EGFRBi-armed autologous activated T cells infused twice a week for 4 weeks for a total of 8 infusions. The doses of the armed ATC will be escalated at the dose levels of 5, 10, 20, and 40 billion armed ATC per infusion. Subcutaneous aldesleukin (300,000IU/m2/day) and Sargramostim (250 ug/m2 twice per week) both starting 3 days before the 1st infusion and ending 7 days after the last dose of armed ATC.
  Other Names: ATC; IL-2; GM-CSF

SUMMARY:
RATIONALE: Giving autologous lymphocytes that have been treated in the laboratory with antibodies may stimulate the immune system to kill tumor cells. Aldesleukin may stimulate the lymphocytes to kill tumor cells. Colony-stimulating factors, such as GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood. Giving laboratory-treated autologous lymphocytes together with aldesleukin and GM-CSF may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of laboratory-treated autologous lymphocytes when given together with aldesleukin and GM-CSF in treating patients with recurrent, refractory, or metastatic advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

Determine the safety and maximum tolerated dose of EGFRBi-armed autologous activated T-cells (ATC) when administered in combination with low-dose aldesleukin and sargramostim (GM-CSF) in patients with recurrent, refractory, or extensive (metastatic) advanced solid tumors.

Secondary

Assess clinical outcome based on tumor responses, overall survival, and progression-free survival.

Monitor changes in sera concentrations of the tumor-associated biomarkers respective of the primary neoplasm (i.e. carcinoembryonic antigen(CEA); prostate specific antigen (PSA); Her2/neu (HER2); etc.) in association with EGFRBi-armed ATC administration throughout the study and at time points thereafter.

Monitor patient sera for human anti-mouse antibodies (HAMA).

Evaluate immune response, which may reflect immune augmentation in response to EGFRBi-armed ATC infusions, in peripheral blood mononuclear cell (PBMC) samples as well as purified immune cell populations.

Investigate proliferation in response to ex vivo stimulation with tumor-specific antigens, sera cytokine profiles (Th1 vs Th2), cytotoxicity of patient PBMC, and interferon gamma ELISPOTS as a surrogate marker for assessing generation of EGFR-specific cytotoxic T-lymphocytes (CTL).

OUTLINE: Peripheral blood mononuclear cells (PBMCs) are collected by 1 or 2 leukaphereses for the generation of activated T cells (ATCs). The PBMCs are activated with OKT3 (anti-CD3) and expanded in aldesleukin for up to 14 days. The ATCs are then armed with EGFRBi.

Patients receive EGFRBi-armed autologous ATCs IV over 30-60 minutes twice weekly for 4 weeks (a total of 8 infusions) in the absence of disease progression or unacceptable toxicity. Patients also receive low-dose aldesleukin subcutaneously (SC) once daily and sargramostim (GM-CSF) SC twice weekly beginning 3 days before the first ATC infusion and continuing for 1 week after the last ATC infusion.

After completion of study therapy, patients are followed periodically.

NOTE: For the purpose of determining safety and maximum tolerated dose of EGFRBi-armed ATC, patients enrolled at each dose level from this study will be combined with patients enrolled at each dose level in RWH 349-32 (NCT00569296): A phase I study of Anti-CD3 x Cetuximab-Armed Activated T Cells, Low Dose IL-2, and GM-CSF for EGFR-Positive, Advanced Non-Small Cell Lung Cancer (NSCLC) to count toward each dose level cohort. A total of three patients enrolled form either of the two trials will be treated at each dose level, but at least one NSCLC patient representative from protocol 349-32 will be enrolled and evaluated at each dose level.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed solid tumor type (ex. Head and Neck Squamous Cell Carcinoma, Colorectal, Pancreatic, Gastric, Esophageal, Renal, Prostate, Breast and Ovarian cancers, etc.); high risk, recurrent, refractory, or metastatic disease after ≥ 1 prior first-line regimen (chemotherapy or radiotherapy)
* Documented EGFR-positive disease (any expression level) by immunohistochemistry (IHC)
* No clinical evidence of active brain metastases; patients with brain metastases are eligible provided they have received definitive radiotherapy or chemotherapy and/or have undergone surgical resection for brain metastases
* No prior hematological malignancy
* Karnofsky performance status (PS) 60-100% OR RCOG PS 0-2
* Life expectancy ≥ 3 months
* Not pregnant or nursing
* Fertile patients must use contraception
* Granulocytes ≥ 1,000/mm3
* Platelet count ≥ 50,000/mm3
* Hemoglobin ≥ 8g/dL
* BUN ≤ 2.0 times normal
* Serum creatinine ≤ 2.0mg/dL
* Bilirubin ≤ 1.5 times normal (with or without liver metastases)
* Hepatitis B surface antigen and HIV negative
* LVEF ≥ 45% at rest by MUGA
* No evidence of depressed left ventricular function
* No other malignancy, except for the following:
* History of curatively treated in situ squamous cell carcinoma or basal cell carinoma of the skin
* History of other curatively treated malignancy (except those with a hematologic origin) for with the patient has remained in complete remission > 5 years after completing therapy (as documented by history, physical exams, tumor markers, and radiology scanning)

Exclusion Criteria

* Serious medical or psychiatric illness that would preclude giving informed consent or receiving intensive treatment
* Recent myocardial infarction (within the past year)
* Current angina/coronary symptoms requiring medications
* Clinical evidence of congestive heart failure requiring medical management (irrespective of MUGA results)
* Systolic blood pressure (BP) ≥ 140 mm Hg or diastolic BP ≥ 90 m Hg; patients with elevated BP must have it controlled by anti-hypertensive medications for at least 7 days prior to the infusion
* Clinical evidence of active brain metastases

Prior/Concurrent Therapy

* More than 4 weeks since prior chemotherapy or radiotherapy
* At least 4 weeks since prior cetuximab or small molecule EGFR-inhibitors including, but not limited to, gefitinib or erlotinib hydrochloride
* No concurrent radiotherapy
* No concurrent steroids except for treatment or adrenal failure, septic shock, or pulmonary toxicity or hormones for non-disease-related conditions(e.g., insulin for diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of EGFRBi-armed autologous activated T-cells | 5 week regimen with 2 month follow up

SECONDARY OUTCOMES:
Determine potential side effects of treating patients with Armed Activated T Cells (ATC) | 5 week regimen with 2 month follow up
Determination of immunologic changes by evaluation of cytokine profiles obtained before and after stimulation with OKT3 in vitro | 5 week regimen with 2 month follow up
Determination of immunologic changes by evaluation of phenotypes of peripheral blood mononuclear cells before and after immunotherapy | 5 week regimen with 2 month follow up
Overall survival | 5 week regimen wtih 2 month follow up
Progression-free survival | 5 week regimen with 2 month follow up
Determination of immunologic changes by evaluation of peripheral blood lymphocytes | 5 week regimen with 2 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Abby Maizel, MD,PhD, Study Chair — Roger William Medical Center
Locations (1):
- Roger Willaims Medical Center, Providence, Rhode Island, United States